CLINICAL TRIAL: NCT03233451
Title: Effect of Psycho-behavioral Intervention on the Depression, Cardiac Function and Quality of Life in Older Adults With Chronic Heart Failure
Brief Title: Psycho-behavioral Intervention for Depression in Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Huali Wang, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-1-4117
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Subjects receive guided psycho-behavioral intervention once a week for 8 weeks. After 8 weeks, the subjects will receive monthly psychological counseling for 7 months.
  Interventions: Behavioral: Psycho-behavioral intervention
- control group (No Intervention): Subjects will receive usual care and be contacted as same frequent as the intervention group.

INTERVENTIONS:
Behavioral: Psycho-behavioral intervention — The psycho-behavioral intervention included 12-week weekly guided psychological intervention (8 modules of behavioral intervention) and 24-week monthly maintenance psychological support.
  Arms: Interventional group

SUMMARY:
The study aims to explore the effectiveness of psycho-behavioral intervention on depressive symptoms among older adults with chronic heart failure. Meanwhile, the effect on cardiac function and quality of life will also be explored.

DETAILED DESCRIPTION:
Depression has been one of the emerging health concerns for older adults, especially for those with chronic heart failure (CHF). It was about 4-5 times more prevalent among patients with CHF than healthy population and independently associated with poor outcome of CHF. As suggested in the clinical management guideline of CHF, it is imperative to create integrative intervention for older adults with CHF, including timely detection and intervention, and ultimately improving the clinical outcome of CHF. However, the approach appropriate for depression intervention among Chinese older adults has yet been developed. This study aims to explore the effectiveness of psycho-behavioral intervention on depression associated with chronic heart failure in old age.

ELIGIBILITY:
Inclusion Criteria:

1. between 60 -85 years old.
2. male or female.
3. Diagnosis with depression as measured with PHQ-9 score of 5 and greater;
4. The subject is diagnosed with chronic heart failure according to their history, symptoms, signs, and adjuvant examinations (eg,echocardiography), in line with the diagnostic criteria for chronic heart failure presented in the China Heart Failure Diagnosis and Treatment Guidelines, with NYHA (New York Heart Association) grade II-III.
5. Reading and writing competency for completing the rating scales.
6. Sufficient physical condition, hearing and vision to ensure the completion of psychological behavior intervention.

Exclusion Criteria:

1. Currently taking antidepressant drugs, and drug dose is unstable.
2. With is a serious risk of suicide, suicide attempts and suicidal behavior (HAMD17 score of 30 or above, or suicide subscale score of 3 and above，or suicide subscale score of MINI of 6 or above).
3. Intact cognitive function with CSI-D score of less than 7.
4. Having other major mental disorders, including Alzheimer's disease, schizophrenia, schizoaffective psychiatric disorders, delusional disorders, undefined psychotic disorders, substance and alcohol abuse
5. Planned heart surgery within 9 months.
6. Unable to comply with psychological intervention due to serious physical conditions -

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
16 Item Quick Inventory of Depressive Symptomatology Self-Report Version | between baseline and week 12
  The primary outcome measure is the response rate of depression from baseline to week 12. The response rate was defined as a 50% or greater score reduction on 16 Item Quick Inventory of Depressive Symptomatology-Self-Report. The total score ranges from 0 to 27, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
16 Item Quick Inventory of Depressive Symptomatology Self-Report Version | between baseline and week 1, 2, 4, 8, 24 and 36
  The severity of depressive symptoms was measured with the 16 Item Quick Inventory of Depressive Symptomatology Self-Report Version. The score ranges from 0 to 27, with higher scores indicating more severe symptoms.
17-Item Hamilton Rating Scale for Depression | between baseline and week 4, 8, 12, 24 and 36
  The severity of depressive symptoms was measured with 17-Item Hamilton Rating Scale for Depression. The 17-item Hamilton Depression Rating Scale produces a total score ranging from 0 (not at all depressed) to 52 (severely depressed).
Beck Depression Inventory II | between baseline and week 1, 2, 4, 8, 12, 24 and 36
  The Beck Depression Inventory II assesses the severity of depression and produces a total score ranging from 0 to 63, with higher scores indicating more severe symptoms.
Geriatric Depression Inventory-Self-Report | between baseline and week 4, 8, 12, 24 and 36
  The Geriatric Depression Inventory-Self-Report assesses the severity of depression and produces a total score ranging from 0 to 12, with higher scores indicating more severe symptoms.
amino-terminal fragment of pro-B-type natriuretic peptide (NT-ProBNP) | between baseline and week 12, and between baseline and week 36
  change of NT-ProBNP level
cardiac function | between baseline and week 12, and between baseline and week 36
  change of ejection fraction as measured with ultrasound cardiogram
Minnesota living with heart failure questionnaire | between baseline and week 4, 8, 12, 24 and 36
  The health-related quality of life was measured by Minnesota Living with Heart Failure Questionnaire.The total score ranges from 0 to 105, with higher scores from best to worst health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Huali Wang, PhD, Principal Investigator — Peking University Institute of Mental Health
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing Chaoyang Third Hospital, Beijing
  - Beijing Fengtai Tieying Hospital, Beijing
  - Beijing Tiancun Community Health Center, Beijing
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
After the results of primary outcome are published, the individual participant data will only be shared anonymously based on request by email to study PI. The team using data should work with the study PI's team on data analysis and publications. The host project should be acknowledged in any submitted working paper, conference presentations and publications.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After the results of primary outcome are published. The data will be available for 2 years.
Access Criteria: Those who are interested in the study should submit a synopsis of research plan for administrative approval by the study committee. Once the data sharing plan is approved by the study committee, the researcher should submit a IRB approval from host institution. When the IRB approval is received, the study committee will ask the data manager to transfer the data for further analysis.

REFERENCES:
- [Derived] Zhang Y, Lv X, Jiang W, Zhu Y, Xu W, Hu Y, Ma W, Sun P, Yang Q, Liang Y, Ren F, Yu X, Wang H. Effectiveness of a telephone-delivered psycho-behavioural intervention on depression in elderly with chronic heart failure: rationale and design of a randomized controlled trial. BMC Psychiatry. 2019 May 27;19(1):161. doi: 10.1186/s12888-019-2135-2. PMID 31132996

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT03233451/SAP_000.pdf